CLINICAL TRIAL: NCT03932266
Title: Endostar Continuous Intravenous Infusion Combined With Induction Chemotherapy and Concurrent Chemoradiotherapy for Locoregionally Advanced Nasopharyngeal Carcinoma (NPC).
Brief Title: Endostar Combined With Induction Chemotherapy and Concurrent Chemoradiotherapy for Locoregional Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Dr. Xia He, Head of radiotherapy department, Jiangsu Cancer Institute & Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endo-Naso-001
Record Dates: First submitted 2017-11-22; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Endostar; Nasopharyngeal Carcinoma; Chemoradiotherapy; Endostatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — endostar protein; Endostatins; Cisplatin; Docetaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Drug: Endostar Drug: Cisplatin Drug: Docetaxel Radiation
  Interventions: Drug: Endostar; Drug: Cisplatin; Drug: Docetaxel; Radiation: Intensity Modulated Radiation Therapy (IMRT)
- Control group (Other): Drug: Cisplatin Drug: Docetaxel Radiation
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Radiation: Intensity Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Drug: Endostar — Endostar, 15 mg/m2, continous intravenous infusion, 3 cycles during induction chemotherapy, 4 cycles during concurrent chemoradiotherapy.
  Other Names: Recombinant human endostatin injection
  Arms: Experimental group
Drug: Cisplatin — Cisplatin, 75 mg/m2, intravenous infusion, 3 cycles during induction chemotherapy; Cisplatin, 80 mg/m2, intravenous infusion, 2 cycles during concurrent chemoradiotherapy.
Drug: Docetaxel — Docetaxel, 75 mg/m2, intravenous infusion, 3 cycles during induction chemotherapy.
Radiation: Intensity Modulated Radiation Therapy (IMRT) — IMRT: 66 Gy, 2-2.2 Gy per fraction, a total of 33 fractions

SUMMARY:
Endostar Continuous Intravenous Infusion Combined With Induction Chemotherapy and Concurrent Chemoradiotherapy for Locoregionally Advanced Nasopharyngeal Carcinoma.

DETAILED DESCRIPTION:
This study was a multicenter, prospective, randomized controlled clinical trial. A set of unified standards were used, including the clinical research program, inclusion criteria, exclusion criteria, chemoradiotherapy regimen and evaluation criteria. A total of 73 patients with pathologically confirmed locoregionally advanced nasopharyngeal carcinoma would be enrolled. Patients were randomly divided into two groups, with 48 patients in the combination group and 25 patients in the control group. The combination group was treated with Induction and Concurrent Chemoradiotherapy combined with Endostar. The control group was treated with Induction and Concurrent Chemoradiotherapy. The short term efficacy and side effects of these treatments would be evaluated. The 1-year, 3-year progression-free survival and overall survival would be analyzed. This data of this study might provide an alternative option for the treatment of Locoregionally advanced nasopharyngeal carcinoma with higher efficacy and low toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or clinically confirmed locally recurrent nasopharyngeal carcinoma;
2. No chemotherapy, immunotherapy, radiotherapy treatment history.
3. No evidence of distant metastasis
4. Eastern Cooperative Oncology Group performance score 0-1
5. Normal bone marrow function: white blood cell count > 3.5 × 109 / L, hemoglobin > 90 g / L and platelet count > 100 × 109 / L.
6. Normal liver function: Alanine aminotransferase (ALT), aspartate aminotransferase (AST) <1.5 times the upper limit of normal (ULN), and alkaline phosphatase (ALP) < 2.5 × ULN
7. Normal renal function: creatinine clearance > 60 ml/min.
8. The patient must be informed of the basic content of the study and sign an informed consent form.

Exclusion Criteria:

1. The pathological type is keratinized squamous cell carcinoma or basal squamous cell carcinoma.
2. Treatment is palliative.
3. A history of malignant tumors, except for well-treated basal cell carcinoma or squamous cell carcinoma and cervical carcinoma in situ.
4. Women during pregnancy or lactation (pregnancy tests should be considered for women of childbearing age; effective contraception should be emphasized during treatment).
5. Previous radiation therapy (except for non-melanoma skin cancer with a previous lesion outside the target area of radiotherapy).
6. Primary and cervical metastatic lesions have received chemotherapy or surgery (except for diagnostic treatment).
7. Having other serious illnesses may result in greater risk or affect the compliance of the trial. For example: kidney disease, chronic hepatitis, control of unsatisfactory diabetes (fasting blood glucose > 1.5 × ULN), and mental illness.
8. A history of severe heart disease, including: cardiac function ≥ standard II, unstable angina, myocardial infarction, arrhythmia - antiarrhythmic drug therapy (except beta-blockers or digoxin), Uncontrollable hypertension.
9. According to the investigator's judgment, there are people with concomitant diseases that seriously endanger the safety of the patient or affect the patient's completion of the study.
10. Patients with a major bleeding tendency in the primary nasopharyngeal tumors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Approximately 36 months
  Progression Free Survival is defined as the time from enrollment to the date of first documented disease progression or death from any cause

SECONDARY OUTCOMES:
objective response rate | 18months
  Complete response (CR)+Partial response (PR) according to RECIST 1.1
overall survival (OS) | Approximately 36 months
  Overall survival was defined as the time from randomization to death from any cause
adverse event (AE) | Approximately 36 months
  adverse event according to NCI-CTCAE (5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Xia He, M.D., Ph.D., Principal Investigator — Jiangsu Cancer Institute & Hospital